CLINICAL TRIAL: NCT01687933
Title: Principal Investigator
Brief Title: The Effect of Virtual Reality Glasses on Labor Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Samira Ebrahimzadeh Zagami, MUMS, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Virtual Reality System
Record Dates: First submitted 2012-08-29; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-08

CONDITIONS: Labor Pain; Anxiety
Keywords: Labor pain; Virtual reality; the first stage of labor; Pain relief; Simulator
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- three-dimensional glasses (Virtual Reality glasses) (Experimental): Women in case group used the glasses for 30 minutes
  Interventions: Device: three-dimensional glasses(manufactor Vuzix,wrap 920)
- usual care (Experimental): Women in control group did not use the glasses.
  Interventions: Other: usual care

INTERVENTIONS:
Device: three-dimensional glasses(manufactor Vuzix,wrap 920) — The samples were randomly allocated to use three-dimensional glasses for 30 minutes in order to reliving labor pain.
  Arms: three-dimensional glasses (Virtual Reality glasses)
Other: usual care — Women in Control group did not use the glasses.
  Arms: usual care

SUMMARY:
There are different medicinal and non medicinal methods to control labor pain. Today, much attention has been on non medicinal methods because of limitations and complications of medical procedures. Virtual reality is a new and promising method of diversion of mind that may have an impact on labor pain. This study was conducted to determine the effect of virtual reality on the first stage of labor pain.

ELIGIBILITY:
Inclusion Criteria:

* Iranian
* low risk pregnancy
* primipara

Exclusion Criteria:

* vision or ear disorders
* History of motion sickness or headaches
* psychological disease or Addiction

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
pain and anxiety | up to 8 months